CLINICAL TRIAL: NCT06931847
Title: SUstaiNable inteRventions and Healthy behavIours for adoleScent Primary prEvention of Cancer With Digital Tools. Study 2: Multiple Behaviour Intervention Platform
Brief Title: SUNRISE Aims to Create a Comprehensive, Engaging, and Sustainable Digital Health Promotion Program That Not Only Addresses Immediate Health Behaviours But Also Instils Lifelong Healthy Habits Among Adolescents. It is a Unique, Digitally Enhanced Program Combining Different Digital Solutions With New
Acronym: SUNRISE_2
Status: Not yet recruiting | Type: Observational
Sponsor: Biobizkaia Health Research Institute (Other Government)
Collaborators: FEDERAZIONE ITALIANA DELLE ASSOCIAZIONI DI VOLONTARIATO IN ONCOLOGIA (Unknown); Hellenic Mediterranean University (Other); University Ghent (Other); University of Zurich (Other); FISABIO (Foundation for the Promotion of Healthcare and Biomedical Research in the Valencian Community) (Unknown); The Oncology Institute "Prof. Dr. Ion Chiricuţă" Cluj-Napoca (Unknown); Cyprus Association of Cancer Patients and Friends (PASYKAF) (Unknown); Alma Mater Europaea University (Unknown)
Responsible Party: Sponsor
Other Study IDs: SUNRISE_Study2; PI2024216 (Other: Comité de Ética de la Investigación con medicamentos de Euskadi (CEIm-E))
Record Dates: First submitted 2024-12-05; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-12

CONDITIONS: Cancer
Keywords: SUNRISE; adolescents; prevention; healthy behaviour; Digital solutions
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: No intervention
- Intervention: SUNRISE program
  Interventions: Other: SUNRISE program

INTERVENTIONS:
Other: SUNRISE program — The program will use several solutions, each focusing on different aspects of health promotion:
  * SmartCoach, a mobile phone-based life-skills training program, focuses on self-management, social skills, and substance use resistance.
  * Social robots and conversational assistants aim to engage students through interactive sessions on health topics like diet and physical activity.
  * Educational and serious games enhance knowledge and resistance to unhealthy food marketing, providing an engaging way to learn about advertising tactics and healthy eating.
  * The influencer campaign tackles nutritional misinformation by using content created by influencers to educate adolescents on detecting and critically evaluating misleading health information.
  * Health and advertisement educational module aims to educate students on recognizing deceptive advertising and making informed choices about their health.
  Groups: Intervention

SUMMARY:
SUNRISE aims to create a comprehensive, engaging, and sustainable digital health promotion program that not only addresses immediate health behaviours but also instills lifelong healthy habits among adolescents. By integrating cutting-edge digital tools with traditional educational settings, SUNRISE seeks to bridge the gap between knowledge and practice, making cancer prevention a tangible and achievable goal for young people. This study represents a significant step towards reducing the future burden of cancer through early and innovative preventive measures.

The SUNRISE project aims to test its interventions on students across eight European countries, including Greece, Switzerland, Slovenia, Spain, Cyprus, Italy, Belgium, and Romania. This study focuses on integrating a unique, digitally enhanced program combining different digital solutions with new methods to change adolescent health behaviour through social media campaigns, social bot platforms, educational games, and health-related advertising content into the school environment, targeting students aged 10 to 19 years.

The program emphasizes inclusivity, ensuring participation from both urban and rural regions and socially disadvantaged groups such as ethnic minorities and migrants. By addressing diverse socio-economic, cultural, and environmental contexts, SUNRISE aspires to create a universally applicable and impactful intervention.

DETAILED DESCRIPTION:
Cancer remains one of the leading causes of death globally, with significant potential for prevention through early adoption of healthy behaviours. Adolescence is a crucial period for establishing such behaviours, and digital interventions offer a promising avenue for promoting sustained health behaviour changes. The SUNRISE project is dedicated to enhancing primary cancer prevention among adolescents in Europe by leveraging innovative digital tools and methodologies.

The Study 2 of the SUNRISE project aims to test its interventions on 4,000 students across eight European countries, including Greece, Switzerland, Slovenia, Spain, Cyprus, Italy, Belgium, and Romania. This study focuses on integrating digitally enhanced programs into the school environment, targeting students aged 10 to 19 years. The program emphasizes in inclusivity, ensuring participation from both urban and rural regions and socially disadvantaged groups such as ethnic minorities and migrants. By addressing diverse socio-economic, cultural, and environmental contexts, SUNRISE aspires to create a universally applicable and impactful intervention.

Adolescence is a period of significant biological, psychological, and social transitions, presenting both opportunities for skill development and risks for harmful behaviours. Substance use often begins during this time, with increased prevalence of alcohol, tobacco, and cannabis consumption as teenagers' age. Furthermore, adolescents are highly susceptible to influences from their social environment, including peers and media. Social media platforms and influencers play a significant role in shaping their attitudes and behaviours, making it essential to leverage these tools to promote healthy behaviours and critical thinking. Schools are ideal settings for preventive interventions due to their accessibility to young people. Platforms like WhatsApp, YouTube, and TikTok offer powerful spaces to reach and engage adolescents, providing interactive functionalities that can impact their health positively. Health behaviour change interventions using social media have shown modest evidence of effectiveness, highlighting the need for further research to target adolescents and ensure the sustainability of behaviour changes in the long term.

SUNRISE sets itself apart from other studies by employing a comprehensive, multi-faceted approach that integrates various digital tools tailored to the specific needs of adolescents. Unlike traditional health promotion programs, which often face challenges in resource allocation and educator support, SUNRISE leverages digital platforms to provide cost-effective, engaging, and personalized interventions. This approach not only makes health information more accessible but also ensures continuous engagement through platforms that adolescents already use for leisure.

The intervention will include a variety of digital tools designed to promote cancer prevention behaviours. These tools will be tailored to the needs of each school through authoring and monitoring platforms, enabling educators to adapt the content and delivery methods. The primary digital solutions include:

* SmartCoach: This mobile-based life-skills training program is designed to prevent substance use by sending tailored messages focusing on self-management, social skills, and substance use resistance. These messages are delivered 2-4 times a week and are integrated with social media platforms to enhance engagement and reach.
* Innovative Social Robots and Conversational Assistants: These tools interact with adolescents through voice commands, offering personalized responses and motivational support. They employ quizzes and persuasive multimedia content to assess and influence health behaviours in areas like diet, physical activity, and advertising literacy.
* Educational and Serious Games: Interactive games designed to improve health knowledge and behaviour. These games are accessible via mobile devices and include scenarios that teach adolescents about the risks of unhealthy food advertising and other health-related topics.
* Influencer Campaigns: Co-created with adolescents, nutrition experts, and influencers, these campaigns aim to combat nutritional misinformation on social media. Influencers will create and share content designed to improve adolescents' understanding and critical evaluation of health information online.
* Health and Advertisement Educational Module: This module uses interactive content such as videos and quizzes to educate adolescents on healthy eating and the tactics used in advertising. It aims to enhance their ability to critically evaluate health messages and make informed decisions.

The implementation of these interventions will be closely monitored and evaluated to assess their effectiveness and sustainability. This will involve statistical analysis of individual outcomes, focus groups, semi-structured interviews with parents, educators, and students, and cost-effectiveness analysis to predict long-term health and economic impacts. The evaluation process is designed to capture a comprehensive picture of how the interventions influence behaviour, well-being, and overall health literacy among adolescents. In addition, PARTICLE.TALK social media platform can collect details of the participants' interaction and its evolution as the study evolves to better support the monitoring and evaluation phases of the study.

SUNRISE aims to create a comprehensive, engaging, and sustainable digital health promotion program that not only addresses immediate health behaviours but also instils lifelong healthy habits among adolescents. By integrating cutting-edge digital tools with traditional educational settings, SUNRISE seeks to bridge the gap between knowledge and practice, making cancer prevention a tangible and achievable goal for young people. This study represents a significant step towards reducing the future burden of cancer through early and innovative preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* Minimum Age: Students must be at least 10 years old at the time of enrolment.
* Devices and Internet Access: Students must have access to an electronic device with Internet connectivity.
* Informed Consent: Students must provide their signed informed consent to participate in the study.
* Parental Consent: Students, when necessary, must obtain and submit signed informed consent from a parent or legal guardian.

Exclusion Criteria:

* Age Restrictions: Students who are younger than 10 years or older than the established age range for participation.
* Consent Issues: Students who have not signed the informed consent form or do not have signed informed consent from their parents or legal guardians.
* Follow-up Limitations: Students who are unable to commit to the follow-up period of at least 18 months or are unlikely to complete the study.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Secondary and upper secondary students between 10 and 19 years old (at time of recruitment), who are freely willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Digitally-Enhanced Program | 18 months
  This will be measured by evaluating the usage and engagement with the intervention, through a in-house authoring and monitoring tool. This tool will include the questionnaires, statistical displays, interactive visualization of data and reporting tools for monitoring and assessment of the intervention outcomes.

SECONDARY OUTCOMES:
Frequency of tobacco cigarette smoking | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Determined by the number of days on which tobacco cigarettes were smoked in the last 30 days
Prevalence and frequency of other nicotine products use | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Determined by the number of days on which other nicotine products, e.g., vape, e-cigarette, e-shisha, snus or nicotine pouches, were consumed in the last 30 days
Prevalence and frequency of cannabis use | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Measured by the number of cannabis (containing THC) consumption days in the preceding 30 days
Prevalence and frequency of alcohol use | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Assessed by the number of alcohol use days in the preceding 30 days
Perceived Stress | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Measured using the 4-item version of the Perceived Stress Scale (PSS-4): The questions in this scale ask about the feelings and thoughts during the last month. In each case, the response represents how often participant felt or thought a certain way.
  Scoring Instructions:
  Total score is determined by adding together the scores of each of the four items. Questions 2 and 3 are reverse coded.
  Questions 1 and 4: 0 = Never; 1 = Almost never; 2 = Sometimes; 3 = Fairly often; 4 = Very often Questions 2 and 3: 4 = Never; 3 = Almost never; 2 = Sometimes; 1 = Fairly often; 0 = Very often Lowest score: 0; Highest score: 16. Higher scores are correlated to more stress.
Social skills | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Assessed utilizing the brief version of the Interpersonal Competence Questionnaire-10 (ICQ-10), which encompasses the following 5 domains: (1) initiation of relationships, (2) negative assertions, (3) disclosure of personal information, (4) emotional support, and (5) conflict management.
  Scoring instructions: Good=4; Fairly good= 3; Rather poor=2; Poor=1. Total score is determined by adding the value of all items and dividing by 2. Maximum value= 20; Minimum value= 5. The higher the score, the higher the interpersonal competence.
Healthy eating habits | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Measured using the WHO/HBSC eating habits questionnaire. Label values: 1 = never, 2 = Less than once a week, 3 = Once a week, 4 = 2-4 days a week, 5 = 5-6 days a week, 6 = Once a day (Every day), 7 = Every Day (more than once).
Physical Activity | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Determined by 2 questions:
  * Over the past 7 days, on how many days were you physically active for a total of at least 60 minutes per day? (0 days - 7 days)
  * Outside school hours: how often do you usually exercise in your free time so much that you get out of breath or sweat? (Every day; 4 to 6 times a week; 2 to 3 times a week; Once a month; Less than once a month; Never)
Health Literacy | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Assessed utilizing the HLS-EU-Q16 Scale that measures health literacy in three domains: health care (seven items), disease prevention (five items) and health promotion (four items). Each question of HLS-EU-Q16 was answered by choosing one response of the available choices: 'very difficult', 'fairly difficult', 'fairly easy' and 'very easy'. Each of the 16 questions were coded according to the following: 'very difficult' = 1 point, 'fairly difficult' = 2 points, 'fairly easy' = 3 points or 'very easy' = 4 points, giving a total of 16-64 scores. The HLS-EU-Q16 manual recommends dichotomising the answers from HLS-EU-Q16 ('very difficult'/'fairly difficult' = 0, 'fairly easy'/'very easy' = 1; total 0-16 scores) and dividing the total scores into three categories ('likely inadequate HL '(0-8 scores), 'likely problematic HL' (9-12 scores) and 'likely sufficient HL' (13-16 scores).
EuroQoL-5D-5L questionnaire | The secondary outcomes will also be assessed at baseline, 6 months, and 18 months follow-up
  Scoring from 0-100 points. 0 points low quality of life 100 high quality of life

CONTACTS AND LOCATIONS:
Locations (8):
- Ghent University (UGENT), Zürich, Belgium
- Cyprus Association of Cancer Patients and Friends (PASYKAF), Nicosia, Cyprus
- Hellenic Mediterranean University (HMU), Heraklion, Greece
- Italian Federation of Voluntary Associations in Oncology (FAVO), Roma, Italy
- Institute of Oncology "Prof dr. Ion Chiricuta" CLUJ NAPOCA (IOCN), Cluj-Napoca, Romania
- Alma Mater Europaea University (AMEU), Maribor, Slovenia
- Foundation for the Promotion of Health and Biomedical Research of the Valencian Community (Fisabio), Valencia, Spain
- Swiss Research Institute for Public Health and Addiction (ISGF), Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Jans S, Spielvogel I, Naderer B, Hudders L. Digital food marketing to children: How an influencer's lifestyle can stimulate healthy food choices among children. Appetite. 2021 Jul 1;162:105182. doi: 10.1016/j.appet.2021.105182. Epub 2021 Mar 3. PMID 33667499
- [Background] Haug S, Paz Castro R, Wenger A, Schaub MP. A Mobile Phone-Based Life-Skills Training Program for Substance Use Prevention Among Adolescents: Cluster-Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Jul 13;9(7):e26951. doi: 10.2196/26951. PMID 34255703
- [Background] Bailey JV, Murray E, Rait G, Mercer CH, Morris RW, Peacock R, Cassell J, Nazareth I. Interactive computer-based interventions for sexual health promotion. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD006483. doi: 10.1002/14651858.CD006483.pub2. PMID 20824850
- [Background] Maher CA, Lewis LK, Ferrar K, Marshall S, De Bourdeaudhuij I, Vandelanotte C. Are health behavior change interventions that use online social networks effective? A systematic review. J Med Internet Res. 2014 Feb 14;16(2):e40. doi: 10.2196/jmir.2952. PMID 24550083
- [Background] O'Keeffe GS, Clarke-Pearson K; Council on Communications and Media. The impact of social media on children, adolescents, and families. Pediatrics. 2011 Apr;127(4):800-4. doi: 10.1542/peds.2011-0054. Epub 2011 Mar 28. PMID 21444588
- [Background] Colditz GA, Wei EK. Preventability of cancer: the relative contributions of biologic and social and physical environmental determinants of cancer mortality. Annu Rev Public Health. 2012 Apr;33:137-56. doi: 10.1146/annurev-publhealth-031811-124627. Epub 2012 Jan 3. PMID 22224878